CLINICAL TRIAL: NCT06084975
Title: Comparison of Outcomes Between Warshaw and Kimura Techniques for Spleen-preserving Minimally Invasive Distal Pancreatectomy: With a Specific Focus on Perioperative Patient Safety
Brief Title: Comparison of Outcomes Between Warshaw and Kimura Techniques for Spleen-preserving Minimally Invasive Distal Pancreatectomy
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Other Study IDs: SP-MIDP
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Distal Pancreatectomy; Spleen Preservation; Postpancreatectomy Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kimura technique (KT): Spleen preservation is accomplished by sparing the splenic vessels.
  Interventions: Procedure: Splenic vessels preservation
- Warshaw technique (WT): Spleen preservation is accomplished by sacrificing the splenic vessels and maintaining vascularity through the preserved short gastric and left gastroepiploic vessels.

INTERVENTIONS:
Procedure: Splenic vessels preservation — preservation the splenic vessels
  Groups: Kimura technique (KT)

SUMMARY:
Spleen-persevering distal pancreatectomy (SP-DP) has been widely advocated as a routine procedure for benign or low-grade malignant tumors in the pancreatic body and tail, especially with a minimally invasive approach. Spleen preservation can be accomplished with Kimura technique (KT) or Warshaw technique (WT) Both of the two techniques were proved to be feasible and efficient. However, the perioperative outcomes and long-term benefits between patients with KT and WT in spleen-persevering minimally invasive distal pancreatectomy (SP-MIDP) remains controversial.

Several small series have reported a slightly higher prevalence of postpancreatectomy hemorrhage (PPH) in patients who undergo KT than those undergo WT. The exposure of splenic vessels to erosive pancreatic juice and the preservation of splenic vessels itself may explain the higher chance of PPH in KT. Larger volume studies are warranted to confirm this finding and to clarify the clinical significance. This study compared the perioperative outcomes between the two spleen-preserving techniques, with a focus on parameters relating to perioperative patient safety. Especially, the incidence and clinical relevance of PPH in SP-MIDP were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis of benign or low-grade malignant pancreas tumors.

Exclusion Criteria:

* incomplete medical records,
* history of previous splenectomy,
* high-grade malignant pancreas tumors,
* conversion to open DP (ODP).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent SP-MIDP at our institution between July 2018 and December 2022 were enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
major complications | Within 30 days of SP-MIDP
  (Clavien-Dindo grade ≥ III)

CONTACTS AND LOCATIONS:
Overall Officials: Liang Tingbo, Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided